CLINICAL TRIAL: NCT03605329
Title: Evaluation of the Severity of Cardiovascular Autonomic Neuropathy in Type 1 Diabetic Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Evaluation of the Severity of Cardiovascular Autonomic Neuropathy in Type 1 Diabetic Patients With OSAS
Acronym: DIADYSAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment rate lower than expected
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF 9801
Record Dates: First submitted 2018-07-09; First posted 2018-07-30 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Sleep Apnea, Obstructive; Diabetes Mellitus, Type 1
Keywords: Sleep Apnea, Obstructive; diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type 1 diabetic patients with OSAS (Other): to explore the severity of NAC in case of OSAS
  Interventions: Other: to explore the severity of NAC in case of OSAS

INTERVENTIONS:
Other: to explore the severity of NAC in case of OSAS — After overnight polysomnography, cardiovascular autonomic neuropathy will be evaluated by different methods: study of HRV, cardiovascular autonomic reflex test (Ewing), measurements of urinary levels of catecholamines and measurements of sweat gland dysfunction using Sudoscan.
  The severity of CAN will be evaluated in T1D patients with moderate to severe OSAS (apnea hypopnea index (IAH) ≥15 / hour) compared to T1D patients with IAH <15 / hour.

SUMMARY:
The links between obstructive sleep apnea syndrome (OSAS) and type 1 diabetes (T1D) are poorly studied. This study proposes to evaluate the severity of cardiovascular autonomic neuropathy (CAN) related to T1D in case of associated OSAS. This issue has significant diagnostic and therapeutic implications because of the increased cardiovascular risk in case of confirmed CAN in T1D patients.

DETAILED DESCRIPTION:
Cardiovascular autonomic neuropathy (CAN) is a common complication of type 1 diabetes (T1D) and is associated with increased cardiovascular risk. Otherwise, some studies have found a high frequence of obstructive sleep apnea syndrome (OSAs) in T1D. Cardiac autonomic modulations are deeply altered in OSAS. The combination of T1D and OSAS could therefore increase the severity of CAN and worsen the cardiovascular prognosis.

The most common method used to explore CAN is the study of heart rate variability (HRV). HRV is a practical, non-invasive and reproducible measure of autonomic nervous system function. HRV abnormalities are a predictor of hypertension and increased mortality in T1D.

Th investigators therefore propose to explore the severity of NAC in case of OSAS associated with T1D, and the hypothesis is that cardiovascular damage is increased in the presence of these two pathologies.

The patients included in this study will be patients with type 1 diabetes diagnosed for more than 5 years.

After overnight polysomnography, cardiovascular autonomic neuropathy will be evaluated by different methods: study of HRV, cardiovascular autonomic reflex test (Ewing), measurements of urinary levels of catecholamines and measurements of sweat gland dysfunction using Sudoscan.

The severity of CAN will be evaluated in T1D patients with moderate to severe OSAS (apnea hypopnea index (IAH) ≥15 / hour) compared to T1D patients with IAH <15 / hour.

Furthermore, glycemic holter will describe the links between glycemic variability, sleep architecture and CAN. Biological oxidative stress assays will improve physiopathological knowledge between T1D, OSAS and CAN. Finally, a 24-hour monitoring of blood pressure will be performed.

An ancillary study is planned to evaluate the evolution of markers of the autonomic nervous system after three months of treatment with CPAP in 15 patients with severe OSAS (AHI ≥30 / hour) having previously participated in the main study. Fifteen patients with IAH <30 / hour will also be reassessed at three months to assess the intra-individual variability of the HRV.

ELIGIBILITY:
Inclusion criteria:

* Type 1 diabetes patients with a diabetes duration of at least 5 years
* Age between 18 and 60 years old.

Exclusion criteria:

* OSAS treated with CPAP
* Chronic alcoholism
* Neuromuscular disease
* Drugs interfering with sinus variability (betablockers, antiarrhythmics, ivabradine), presence of pacemaker
* Pregant woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
study of heart rate variability (HRV) | day 1
  heart rate variability (LF/HF ratio) in type 1 diabetic patients with sleep apnea syndrome (AHI>15/h) in comparison with T1D patients with AHI <15/hour.

SECONDARY OUTCOMES:
Evaluation of the severity of CAN | day 1
  measurements of urinary levels of catecholamines
measurements of sweat gland dysfunction | day 1
  Sudoscan
Characterization of the sleep architecture of T1D patients | day 1
  overnight polysomnography
monitoring of blood pressure | day 1
  a 24-hour monitoring of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: François Bughin, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France